CLINICAL TRIAL: NCT01010308
Title: Nadolol for Proliferating Infantile Hemangiomas: A Prospective Open Label Study With a Historical Control
Brief Title: Nadolol for Proliferating Infantile Hemangiomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Elena Pope, Staff Physician, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000014079
Record Dates: First submitted 2009-11-08; First posted 2009-11-10 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Infantile Hemangioma
Keywords: infantile hemangioma; nadolol
MeSH Terms: conditions — Hemangioma, Capillary | interventions — Nadolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention Group: (Experimental): The patients in this study are infants aged 1 month to 1 year of age with head and neck hemangiomas currently causing /or with impending function loss (e.g. vision, airway obstruction, feeding, etc), or hemangiomas currently causing/or with potential for facial disfigurement
  Infants aged 1 month to 1 year of age with head and neck hemangiomas that received treatment with systemic propranolol in the past 2 years as a control group
  Interventions: Drug: Nadolol
- Historical control group (No Intervention): Ten infants (1-12 months of age) treated with propranolol will be identified from a Dermatology Database. Patients will be considered as controls if they were treated with propranolol before 1 year of age and had digital photography documentation of their hemangioma.
- Angiogenesis marker control group (No Intervention): The angiogenesis marker control group will consist of 6 -10 patients seen in the Dermatology clinic for conditions other than IH and not receiving corticosteroids or beta blockers.

INTERVENTIONS:
Drug: Nadolol — Nadolol will be administered orally at home starting at 0.5 mg/kg/day divided into 2 doses. Weekly, if BP and heart rate are acceptable, the dose will be increased by 0.5 mg/kg/day up to 2 mg/kg/day.
  Arms: Intervention Group:

SUMMARY:
The purpose of this study is to explore the efficacy and safety of Nadolol in hemangiomas of infancy.

The secondary objective is to assess the feasibility of conducting a randomized controlled trial comparing nadolol with corticosteroids and propranolol.

DETAILED DESCRIPTION:
Systemic corticosteroids are currently the most frequent used medication for treatment of problematic infantile hemangiomas (IH's). Since June 2008, systemic propranolol has been an important addition to the therapeutic options for problematic IH, allowing decreased dependence on the systemic corticosteroids. So far, we have found excellent response with propranolol with minimal short-term side effects. Studies, which compared nadolol and propranolol in children with other conditions, suggest that nadolol is safer and more efficacious than propranolol. In addition, it has better dosing schedules and less central nervous system (CNS) penetration, making it suitable even for patients with suspected or proven PHACES syndrome.

ELIGIBILITY:
Inclusion Criteria:

Intervention Group

* Infants aged 1 month to 1 year of age with head and neck hemangiomas currently causing /or with impending function loss (e.g. vision, airway obstruction, feeding, etc), or hemangiomas currently causing/or with potential for facial disfigurement.

Historical Control Group

* Infants aged 1 month to 1 year of age with head and neck hemangiomas that received treatment with systemic propranolol in the past 2 years

Angiogenesis Marker Control Group

* Infants aged 1 month to 1 year attending dermatology clinic

Exclusion Criteria:

Intervention Group

* Patients with PHACES syndrome (proven) or suspected PHACES (plaque like hemangioma awaiting imaging).
* Children with history of hypersensitivity to beta blockers
* Children with personal history or family history of a first degree relative with asthma
* Children with known renal impairment
* Children with known cardiac conditions which may predispose to heart blocks
* Personal history of hypoglycemia
* Children on medications that may interact with beta blockers

Historical Control Group:

* No digital photography available documenting IHs progression

Angiogenesis Marker Control Group:

* Children with IH
* Children on beta blocker or systemic corticosteroids

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with at least 75% improvement in the extent of the hemangioma | Baseline, 6months

SECONDARY OUTCOMES:
The proportion of subjects with at least 50% improvement in the extent of the hemangiomas | Baseline and 6 months
  The proportion of subjects with at least 50% improvement in the extent of the hemangiomas
The percentage of patients with >75% improvement in the Nadolol group compared to a historical cohort of patients receiving propranolol. | 6 months
  The percentage of patients with >75% improvement in the Nadolol group compared to a historical cohort of patients receiving propranolol.
The correlation between the changes in the levels of angiogenesis markers and clinical response to treatment. | 6 months
  The correlation between the changes in the levels of angiogenesis markers and clinical response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Pope, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada